CLINICAL TRIAL: NCT00317486
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Tracleer (Bosentan) on Oxygen Saturation and Cardiac Hemodynamics in Patients With Pulmonary Arterial Hypertension Related to Eisenmenger Physiology
Brief Title: Effects of Tracleer (Bosentan) on Pulmonary Arterial Hypertension Related to Eisenmenger Physiology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-052-405
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension Related to Eisenmenger Physiology
Keywords: pulmonary arterial hypertension; Eisenmenger physiology; bosentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

INTERVENTIONS:
Drug: bosentan

SUMMARY:
This study evaluates the effects of bosentan on oxygen saturation, hemodynamics and exercise capacity in patients with pulmonary arterial hypertension related to Eisenmenger physiology. Patients receive bosentan or placebo for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 12 years with a body weight at least 40 kg (inclusive) and with a functional class III (1998 WHO classification).
2. Patients with pulmonary arterial hypertension related to Eisenmenger physiology echocardiographically established as atrial septal defect at least 2 cm effective diameter and/or ventricular septal defect at least 1 cm effective diameter; PAH confirmed via cardiac catheterization: mean pulmonary arterial pressure >25 mm Hg, pulmonary capillary wedge pressure <15 mm Hg and pulmonary vascular resistance >3 mm Hg/l/min.
3. Patients with documented oxygen saturation up to 90%, and >70% (at rest, with room air).
4. Patients able to perform a 6-minute walk test at least 150 m, and up to 450 m.
5. Patients stable for at least 3 months prior to screening.
6. Bosentan naïve patients.
7. Female patients who are surgically sterile, postmenopausal or have documented infertility.
8. Female patients of childbearing potential using one of the following methods of contraception: Barrier-type devices (e.g., condom, diaphragm) used ONLY in combination with a spermicide. A double-barrier method is recommended; intrauterine devices (IUDs); oral or implanted contraceptives, if used in combination with a barrier method.
9. Patients providing written informed consent.

Exclusion Criteria:

1. Pregnant patients, nursing mothers.
2. Patients with left ventricular dysfunction (ejection fraction <40%).
3. Patients with restrictive lung disease (TLC<70% predicted); obstructive lung disease (FEV1<70% predicted, with FEV1/FVC<60%)
4. Patients with systolic blood pressure < 85 mm Hg.
5. Patients with other conditions that may affect the ability to perform a 6-minute walk test.
6. Patients unable to provide informed consent and comply with the patient protocol.
7. Patients with known coronary arterial disease.
8. Patients with serum creatinine >125 µM/l.
9. Patients with iron deficiency (serum ferritin <10 ng/ml) unless corrected by iron supplement.
10. Patients with hemoglobin or hematocrit that is more than 30% below the normal range (patients with secondary polycythemia are permitted).
11. Patients with AST and/or ALT values greater than 3 times the upper limit of normal.
12. Patients who have started or stopped treatment for PAH within one month of screening, excluding anticoagulation.
13. Patients who are receiving glyburide (glibenclamide), cyclosporine A or tacrolimus at inclusion or are expected to receive any of these drugs during the study.
14. Patients who are receiving vasodilators including, but not limited to epoprostenol or prostacyclin analogues, or are expected to receive any of these drugs during the study.
15. Patients active on organ transplant lists.
16. Patients taking phosphodiesterase inhibitors or endothelin receptor antagonists (other than bosentan) or any other investigational drugs/devices.
17. Patients with planned surgical intervention during the study period.
18. Cardiac catheterization-specific exclusion criteria:

    1. Patients who cannot safely have catheterization performed as indicated.
    2. Patients in whom shunting is not at the atrial or ventricular level.
    3. Patients with nonequal pulmonary venous desaturation that theoretically cannot be corrected with administration of 100% non-rebreather-supplied oxygen.
    4. Patients with nonpulsatile pulmonary blood flow, or with multiple sources of pulmonary blood flow.
    5. Patients with discontinuous pulmonary arteries, peripheral pulmonary arterial or venous stenosis > 25% size of native PA or creating unequal bilateral PA mean pressures, PA band with gradient > 20 mm Hg, tetralogy of fallot/pulmonary atresia, VSD/pulmonary atresia, DORV/pulmonary atresia, truncus arteriosus, scimitar syndrome.
    6. Patients where SVC sampling cannot be performed, or where SVC sampling may be contaminated
    7. Patients with ductus arteriosus.
    8. Patients with mitral or pulmonary venous stenosis, intracavitary LV outflow obstruction, sub, valvar or supravalvar aortic stenosis or aortic coarctation.
    9. Patients with <10 indexed Wood units, greater than moderate mitral regurgitation, mean pulmonary venous pressure > 16 mm Hg, pulmonary venous "v" waves > 20 mm Hg, systemic ventricular end-diastolic pressure > 16 mm Hg; patients with recognized extracardiac systemic venous collaterals to the pulmonary venous circulation, patients with recognized hepatic wedge pressure-inferior vena cava pressure gradient > 12 mm Hg.
    10. Patients (during catheterization) with uncorrectable hypercarbia with pCO2 >55 mm Hg; patients with uncorrectable acidemia with pH <7.34; patients in active pain or distress; unconscious or mechanically ventilated patients; patients with unstable systemic or pulmonary blood flow; systemic arterial or pulmonary artery pressures or hematocrit (change of > 25% during catheterization); unstable cardiac rhythm dissimilar to baseline cardiac rhythm during physical examination assessments for the entire duration of the catheterization excepting nonsustained arrhythmia; patients with documented or recognized air embolism, hemorrhage, cardiac, cerebral or peripheral organ ischemia occurring during or immediately preceding the catheterization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-09; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 16 in oxygen saturation at rest with room air
Change from baseline to Week 16 in indexed pulmonary vascular resistance

SECONDARY OUTCOMES:
Changes from baseline to Week 16 in cardiac hemodynamics